CLINICAL TRIAL: NCT00406783
Title: Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter/Multinational, Efficacy and Safety Study of Desloratadine 5 mg in the Treatment of Subjects With Allergic Rhinitis Who Meet the Criteria for Intermittent Allergic Rhinitis (IAR)
Brief Title: Study for the Treatment of Intermittent Allergic Rhinitis With Desloratadine (Study P04683)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04683
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Results first posted 2009-03-06 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial
Keywords: Allergic Rhinitis; Intermittent Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-mg Desloratadine tablet (Experimental)
  Interventions: Drug: 5-mg Desloratadine
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-mg Desloratadine — 5-mg Desloratadine tablet, once daily for 15 days
  Other Names: SCH 34117, Aerius
  Arms: 5-mg Desloratadine tablet
Drug: Placebo — Placebo tablet, once daily for 15 days
  Arms: Placebo tablet

SUMMARY:
This study will investigate the effectiveness of desloratadine in treating subjects with allergic rhinitis (AR) who meet the criteria for intermittent allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

The subject must meet ALL of the criteria listed below for entry:

* For this study, the diagnosis of IAR is not based solely on the current episode of AR. Subjects must have at least a 2 year history of AR consistent with IAR (defined as symptoms of allergic rhinitis present less than four days per week or for less than four consecutive weeks per year); the current episode can count as the second year.
* Subjects must be 12 years of age and older, of either sex and of any race.
* At the Run-In Visit, subjects must be sufficiently symptomatic, with a T5SS 12-hour AM-PRIOR (reflective) symptoms severity score of at least 6.
* In order for a subject to qualify at the Baseline Visit, the sum of the daily averages of the diary recordings of the 12-hour AM PRIOR + PM-PRIOR (reflective) T5SS collected during Days -4 to -1 and the AM PRIOR T5SS on the morning of the Baseline Visit (Day 1) must be >= 30.
* Subjects must have a positive skin-prick test at screening to one or more allergens in the GA2LEN (or the usually used local) panel of seasonal and perennial allergens. Subjects must demonstrate an antigen-induced skin prick wheal at least 3 mm in diameter greater than diluent control. The positive tests must include the allergen(s) prevalent while this study is active.
* Subjects must be free of any clinically significant disease, other than IAR, which would interfere with the study evaluations.
* Subjects, or parents/legal guardians, must give written informed consent. Subjects must be able to adhere to dose and visit schedules and meet study requirements.
* In females of childbearing potential, the urine pregnancy test (hCG) must be negative at the Screening Visit.
* Nonsterile or premenopausal female subjects must be using a medically accepted method of birth control, that is, oral contraceptive, hormonal implant, medically prescribed intrauterine device (IUD), or depot injectable during the entire study. A female subject who is not currently sexually active must agree and consent to use one of the above-mentioned methods, if she becomes sexually active while participating in the study. A female subject who is not of childbearing potential must have a medical record of being surgically sterile (for example, hysterectomy and tubal ligation), or be at least 1 year postmenopausal.

Exclusion Criteria:

The subject will be excluded from entry if ANY of the criteria listed below are met:

* Subjects with a history of anaphylaxis and/or severe local reaction(s) to skin testing with allergens.
* Subjects with intolerable symptoms that would make participating in the study unbearable.
* Subjects who have had an upper respiratory tract or sinus infection that required antibiotic therapy, and have not had at least a 14-day washout prior to the run-in period, or who have had a viral upper respiratory infection within 7 days prior to screening.
* Subjects with asthma who require chronic use of inhaled or systemic corticosteroids.
* Subjects with current or a history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* Subjects on immunotherapy (desensitization therapy) unless on a regular maintenance schedule prior to Visit 1 and staying on this schedule for the remainder of the study.
* Subjects who, in the opinion of the investigator, are dependent on nasal, oral or ocular decongestants, nasal topical antihistamines or nasal steroids.
* Subjects who have used any drug or device in an investigational protocol in the 30 days prior to Visit 1.
* Female subjects who are pregnant or nursing.
* Subjects with a history of hypersensitivity to the study drug or to their excipients or known to not tolerate any antihistamines.
* Subject is a member of the Investigational Study Staff (currently involved with this study) or a member of the staff's family.
* Subjects with current evidence of clinically significant hematopoietic, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disease, or other diseases that preclude the subject's participation in the study.
* Subjects whose ability to provide informed consent is compromised.
* Subjects with a history of noncompliance with medications or treatment protocols.
* Subjects with rhinitis medicamentosa.
* Subjects who have, in the opinion of the investigator or designee, clinically significant nasal structural abnormalities, including large nasal polyps or marked septum deviation, that significantly interferes with nasal air flow.
* Subjects who have not observed the medication washout times outlined in the protocol prior to Visit 2.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bousquet J, Bachert C, Canonica GW, Mullol J, Van Cauwenberge P, Bindslev Jensen C, Fokkens WJ, Ring J, Keith P, Lorber R, Zuberbier T; ACCEPT-1 study group. Efficacy of desloratadine in intermittent allergic rhinitis: a GA(2)LEN study. Allergy. 2009 Oct;64(10):1516-1523. doi: 10.1111/j.1398-9995.2009.02115.x. Epub 2009 Jul 14. PMID 19624554

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-mg Desloratadine Tablet: 5 mg desloratadine tablet, once daily for 15 days
- Placebo Tablet: placebo tablet, once daily for 15 days
Period: Overall Study
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Started | 276 | 271
Completed | 262 | 256
Not Completed | 14 | 15
Not completed — Adverse Event | 4 | 4
Not completed — Treatment Failure | 2 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Protocol Violation | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet | Total
Number analyzed (Participants) | 276 | 271 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (12.0) | 34.6 (12.8) | 34.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 164 | 318
  Male | 122 | 107 | 229

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in the 12-hour AM/PM-PRIOR (Reflective) Total 5 Symptom Score (T5SS) From Subject Daily Diaries Averaged Over Treatment Days 1 to 15
Description: AM/PM is the average of separate morning (AM) and evening (PM) evaluations. T5SS = the sum of the individual scores for nasal congestion/stuffiness, sneezing, rhinorrhea/nasal discharge, nasal pruritis, and ocular pruritis. Each individual symptom/sign was scored from 0 (none) to 3 (severe).
Time Frame: 15 days
Population: Last Observation Carried Forward (LOCF) to the final visit. All randomized subjects with a non-missing baseline and at least some post-baseline data were included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 271 | 265
scores on a scale | -3.01 (0.21) | -2.13 (0.2)
Statistical Analysis 1: Comparison: 5-mg Desloratadine Tablet vs Placebo Tablet; Test type: Superiority or Other; p < 0.001, ANOVA

2. Secondary Outcome: Change From Baseline in the Rhinoconjunctivitis Quality of Life Questionnaire-Standardized Version (RQLQ-S) at the Final Visit
Description: The RQLQ-S questionnaire consists of 28 questions grouped into 7 domains. Each question is scored on a scale of 0 (not troubled with symptoms) to 6 (extremely troubled with symptoms). The total RQLQ-S score is the average score of the 28 questions which consisted of a total of 7 domains.
Time Frame: 15 days
Population: Last Observation Carried Forward (LOCF) to the final visit. The RQLQ-S was only completed for subjects >=18 years of age and where available in the local language.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 250 | 248
scores on a scale | -1.1 (0.1) | -0.73 (0.1)
Statistical Analysis 1: Comparison: 5-mg Desloratadine Tablet vs Placebo Tablet; Test type: Superiority or Other; p < 0.001, ANOVA

3. Other Pre Specified Outcome: Total 5 Symptom Score (T5SS) - Average AM/PM PRIOR (Reflective) 12 Hours Diary: BASELINE
Description: as for outcome 1
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 271 | 265
scores on a scale | 8.5 (0.14) | 8.33 (0.14)

4. Other Pre Specified Outcome: Rhinoconjunctivitis Quality of Life Questionnaire-Standardized Version (RQLQ-S: BASELINE
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Number analyzed (Participants) | 250 | 248
scores on a scale | 2.96 (0.08) | 2.80 (0.08)

ADVERSE EVENTS:
Description: Subjects were questioned and/or examined by the investigator for evidence of adverse events. The questioning of subjects with regard to the possible occurrence of adverse events were to be generalized such as, "How have you been feeling since your last visit?"
Arm/Group | 5-mg Desloratadine Tablet | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/276 | 0/271
Other Adverse Events (participants affected / at risk) | 18/276 | 17/271
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Desloratadine Tablet (N=276) | Placebo Tablet (N=271)
Headache (Nervous system disorders) | 18 (23) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide sponsor w/ review copies of abstracts or manuscripts for publication that report any results of the study, 45 days before submission for publication or presentation. The sponsor shall have the right to review/comment on the material. If the parties disagree about the appropriateness of the material, PI must meet with sponsor's representatives before submission for publication, for the purpose of making good faith efforts to discuss and resolve any issues of disagreement.